CLINICAL TRIAL: NCT01481948
Title: Using Technology to Prevent Obesity Among African American Girls
Brief Title: Food, Fun, & Fitness Internet Program for Girls: Outcome Evaluation
Acronym: FFFIPG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Deborah Thompson, Associate Professor of Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-27505; R01MD005814 (NIH)
Record Dates: First submitted 2011-11-21; First posted 2011-11-30 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
Keywords: physical activity; fruit and vegetable; water; girls; African American; online
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- story plus behaviorial procedures (Experimental): The girls randomized to this arm of the study will view an interactive story about 6 8-10 year old African American girls who seek to find clues to solve a mystery about the town in which they live. The episodes will contain information about healthy nutrition and physical activity, as well as basic information about physical activity and kitchen safety tips, developmentally appropriate recipes, and portion sizes. Girls randomized to this arm of the study will also engage in key behavior change procedures, such as goal setting, problem solving, and self monitoring.
  Interventions: Behavioral: Food, Fun, & Fitness Internet Program for Girls
- story only (Active Comparator): The girls randomized to this arm of the study will view an interactive story about 6 8-10 year old African American girls who seek to find clues to solve a mystery about the town in which they live. The episodes will contain information about healthy nutrition and physical activity, as well as basic information about physical activity and kitchen safety tips, developmentally appropriate recipes, and portion sizes. Girls randomized to this arm of the study will not engage in key behavior change procedures, such as goal setting, problem solving, and self monitoring.
  Interventions: Behavioral: Food, Fun, & Fitness Internet Program for Girls
- Wait list control (No Intervention): This group will participate in data collection only; after the 3rd data collection point, they will be given access to the intervention

INTERVENTIONS:
Behavioral: Food, Fun, & Fitness Internet Program for Girls — This is an 8 episode intervention, delivered entirely over the internet. Each episode, girls will view an interactive story in which 6 8-10 year old African American characters attempt to solve a mystery about their town. The online program will include information about healthy nutrition (i.e., consuming more fruit, vegetables, water) and physical activity. There will be two groups; one group (the experimental group) will view the interactive story and participate in key behavior change procedures, such as personal goal setting, problem solving, and self monitoring activities. The second group (the active comparator group) will view the online stories but will not engage in key behavior change procedures.
  Arms: story only; story plus behaviorial procedures

SUMMARY:
The purpose of this project is to reduce health disparities in obesity risk among 8-10 year old African American girls using a culturally sensitive and developmentally appropriate internet-based program with no face-to-face interaction. This study will conduct an outcome evaluation to test short and longer term effects on obesity risk.

DETAILED DESCRIPTION:
This research will conduct an outcome evaluation on a promising web based obesity prevention program for 8-10 year old African American girls. A pilot study with 80 girls established its feasibility: recruitment goals were met; attrition rates were < 10%; logon rates to the online program were 74.5%; and statistically significant increases in fruit and vegetable consumption and time spent being physically active were observed. The outcome evaluation will recruit 400 child-parent pairs to examine short and longer term effects of the program on obesity risk. It will also conduct mediation analyses to examine pathways of effect. At the end of the study, the web based program will be hosted on the CNRC web site. Although the use of the internet as a method for changing health behavior is not new, the use of an internet program alone, with no face to face interaction, is novel. This is one of the first programs to attempt this, particularly in an at-risk population.

ELIGIBILITY:
Inclusion Criteria:

* 8-10 years old
* healthy
* African American
* parent willing to participate in data collection
* internet access
* personal email address

Exclusion Criteria:

* mental, physical, or medical conditions that limit fruit-vegetable consumption, physical activity, or ability to fully participate in the program and/or complete baseline and post assessment data collection
* taking medications that influence dietary behaviors, appetite, and/or physical activity

Ages: 8 Years to 10 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 342 (Actual)
Dates: Start 2012-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Body mass index percentile | 6 months
  height and weight will be used to calculate BMI percentile

SECONDARY OUTCOMES:
fruit and vegetable consumption | 3 months
  dietitian-assisted dietary recalls will be collected using the NDSR system; 2 recalls will be collected (1 week day and 1 weekend day)
physical activity | 3 months
  Accelerometers will be used to assess physical activity at each time point
self efficacy | 3 months
  Standard measures will be used to assess fruit, vegetable, water, and physical activity self efficacy
home availability | 3 months
  standard measures will be used to assess fruit, vegetable, and physical activity equipment home availability
asking behaviors | 3 months
  standard measures will be used to assess child fruit, vegetable, water, and physical activity asking behaviors
fruit and vegetable consumption | 6 months
  dietitian-assisted dietary recalls will be collected using the NDSR system; 2 recalls will be collected at each time point (1 week day and 1 weekend day)
physical activity | 6 months
  Accelerometers will be used to assess physical activity
self efficacy | 6 months
  standard measures will be used to assess fruit, vegetable, water, and physical activity self efficacy
home availability | 6 months
  standard measures will be used to assess fruit, vegetable, and physical activity equipment home availability
asking behaviors | 6 months
  standard measures will be used to assess child fruit, vegetable, water, and physical activity asking behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Deborah I Thompson, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] Callender C, Liu Y, Moore CE, Thompson D. The baseline characteristics of parents and African American girls in an online obesity prevention program: A feasibility study. Prev Med Rep. 2017 May 19;7:110-115. doi: 10.1016/j.pmedr.2017.05.011. eCollection 2017 Sep. PMID 28652960
- [Derived] Thompson D, Mahabir R, Bhatt R, Boutte C, Cantu D, Vazquez I, Callender C, Cullen K, Baranowski T, Liu Y, Walker C, Buday R. Butterfly Girls; promoting healthy diet and physical activity to young African American girls online: rationale and design. BMC Public Health. 2013 Aug 2;13:709. doi: 10.1186/1471-2458-13-709. PMID 23915235